CLINICAL TRIAL: NCT02559193
Title: Medication Interactions to Detect Adverse Situations
Brief Title: Pharmacogenetic Testing for Medication Management.
Status: Withdrawn | Type: Observational
Why Stopped: Loss of funding for the continuation of the Study
Sponsor: First Vitals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MIDAS
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Medication Management
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment.: Data collection only trial design.
  Interventions: Other: Observational study, data collection only trial.

INTERVENTIONS:
Other: Observational study, data collection only trial. — Data collection only trial design.

SUMMARY:
The Study is a single-arm prospective trial of patients receiving at least one medication with a known association between genetics and drug metabolism. All patients will undergo genetic testing as determined by their treating physician. The specific genes tested will, in general, be based upon the drugs the patients are taking or those that the patient's treating physician is considering as potential substitutes for current medications.

DETAILED DESCRIPTION:
In this data collection only trial design, the PGx test is not a protocol-specified procedure. Rather, patients are eligible if they have undergone PGx testing within the last 90 days. Thus, PGx testing will not be performed solely for inclusion in this clinical research initiative.

ELIGIBILITY:
Inclusion Criteria:

1. Patient underwent PGx testing for alleles appropriate to the target drugs within the prior 90 days ("index PGx test");
2. Male or female patients 18 years or older who have given their written Informed Consent to participate in a Clinical Study based on voluntary agreement a through explanation of the patient's participation is provided to them. Patients must have adequate reading and writing abilities such that they can comprehend and answer the questions on the patient- completed assessments and Informed Consent Form;
3. Patient was receiving at least one medication known to be associated with allelic variation at the time of the index PGx test), including over-the-counter medications;

5. Patient has a history of at least one TDAE over the 12-month period preceding receipt of PGx test results, or has experienced inadequate efficacy from a target drug and receiving medical coverage through a private insurance.

Exclusion Criteria:

1. Patient is currently hospitalized;
2. Patient's medical and medication history is unavailable over the 90-day period preceding the receipt of PGx testing;
3. Patient is unable to provide an accurate history due to mental incapacity;
4. Patient is known to have undergone prior PGx testing for genes specific to the target drug(s), exclusive of the PGx test relating to this Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Study will include male or female patients 18 years of or older who are receiving at least one medication with metabolism known to depend on genetic variation and have the PGx test already performed. The patient must also meet the inclusion/ exclusion criteria established by the protocol.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the Study is the binary occurrence of meaningful change in drug regimen. | 90-day period following receipt of PGx test results

CONTACTS AND LOCATIONS:
Overall Officials: Ernie Lee, CHRS, Study Director — First Vitals LLC